CLINICAL TRIAL: NCT02359344
Title: A Randomized, Double-blind, Placebo Controlled, Two Period Crossover Study to Investigate the Pharmacokinetics, Tolerability and Cognitive Effects of an Oral Dose Regimen of 150mg Tid CNV1014802 in Healthy Young Versus Elderly Male and Female Subjects
Brief Title: PK & Tolerability of CNV1014802 in Young and Elderly Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1014802/101; 2014-004980-19 (EudraCT Number)
Record Dates: First submitted 2015-02-02; First posted 2015-02-10 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — vixotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CNV1014802 (Experimental): CNV1014802 150mg three times a day (tid) 7 days plus a single dose on day 8
  Interventions: Drug: CNV1014802
- Placebo (Placebo Comparator): Placebo tid 7 days plus a single dose on day 8
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CNV1014802
  Other Names: BIIB074
  Arms: CNV1014802
Drug: Placebo
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo controlled, two period crossover study to investigate the pharmacokinetics, tolerability and cognitive effects of 8 days dosing of CNV1014802 in healthy young versus elderly male and female subjects. Treatment periods will be separated by 13 days. The primary outcome measures are pharmacokinetics (PK) and tolerability.

DETAILED DESCRIPTION:
This study was previously posted by Convergence Pharmaceuticals, Ltd., which has been acquired by Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male and female over 18 years using acceptable methods of contraception

Key Exclusion Criteria:

* Positive pre-study HIV, Hepatitis B surface antigen or positive Hepatitis C antibody
* History or evidence of alcohol or drug abuse
* Pregnant or lactating females
* Participation in a clinical trial within 3 months or the current study or exposure to more than four new chemical entities within 12 months.
* Use of prohibited concomitant medication
* History or presence of any clinically significant abnormality in vital signs / ECG / laboratory tests, or have any medical or psychiatric condition, which, in the opinion of the Investigator may interfere with the study procedures or compromise subject safety.
* Relevant history of a suicide attempt or suicidal behavior

Note: Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2015-04-20 (Actual); Study Completion 2015-04-20 (Actual)

PRIMARY OUTCOMES:
Maximum Concentration | 9 days
Area under the concentration curve | 9 days
Minimum concentration | 9 days
Frequency of adverse events | 9 days
Change in vital signs compared to baseline | 9 days
Change in 12-lead ECG parameters compared to baseline | 9 days
Change in safety lab parameters compared to baseline | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Parexel International, London, United Kingdom